CLINICAL TRIAL: NCT05220202
Title: MOTIVATE to Improve Outcomes for Older Veterans With Musculoskeletal Pain and Depression
Acronym: MOTIVATE_IIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Dallas VA Medical Center (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 20-256; IRB # 1672072 (Other: Dallas VA Medical Center)
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Chronic Back Pain; Depression; Aging; Musculoskeletal Pain
Keywords: Chronic Back Pain; Depression; Veterans; Aging; Musculoskeletal Pain
MeSH Terms: conditions — Depression; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: This Randomized Clinical Trial will randomize to either MOTIVATE or a waitlist control
Who Masked: Outcomes Assessor
Masking Description: The research staff conducting outcome assessments will be blinded to whether the subject is in active or waitlist group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Waitlist Control Group (No Intervention): The waitlist control group will continue with usual care management of musculoskeletal pain and depression. All participants, regardless of what group they have been assigned to will undergo several outcome assessments (pre-screening, baseline, midpoint, final assessments) conducted by a blinded research assistant. Subjects randomized to the waitlist control group will be offered the intervention once they have completed the end outcomes assessment.
- Behavior Intervention Group (MOTIVATE) (Experimental): For participants assigned to the intervention arm, trained health coaches will deliver the 8 session intervention via telephone. MOTIVATE users motivational interviewing techniques, values elicitation and physical activity based goal setting. All participants, regardless of what group they have been assigned to will undergo several outcome assessments (pre-screening, baseline, midpoint, final assessments) conducted by a blinded research assistant.
  Interventions: Behavioral: Behavioral Intervention Group (MOTIVATE)

INTERVENTIONS:
Behavioral: Behavioral Intervention Group (MOTIVATE) — Behavioral: Behavioral Intervention Group (MOTIVATE) The behavioral intervention is designed for older Veterans with musculoskeletal pain and depression and will include 8 individual telephone sessions delivered by health coaches (for up to 5 months total), accounting for additional time between sessions (if needed).
  Other Names: MOTIVATE
  Arms: Behavior Intervention Group (MOTIVATE)

SUMMARY:
The proposed study seeks to evaluate effectiveness, implementation processes, and cost of MOTIVATE among older Veterans with chronic musculoskeletal (MSK) pain and comorbid depressive symptoms.

DETAILED DESCRIPTION:
Investigators will conduct a randomized controlled trial (RCT) at two large VA facilities, to establish the effectiveness and scalability of MOTIVATE, a remotely delivered behavioral intervention for older Veterans with comorbid musculoskeletal (MSK) pain and depressive symptoms. The central hypothesis is that MOTIVATE will improve important patient-centered outcomes among older Veterans with co-occurring MSK pain and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 and older
* English- speaking
* Self-reported MSK pain (include cLBP +/- radiating symptoms, OA, fibromyalgia) on most days for the past 3 months that interferes with daily activities
* Pain intensity that is 4+/10 on the numerical pain rating scale
* Pain interference threshold 5+ on PEG-3
* Depressive symptoms, 10+ on PHQ-9
* Capable of participating in home-based activity
* Interested in participating in a non-pharmacologic program

Exclusion Criteria:

* Aged 59 or less
* No telephone
* Not English speaking
* Unwilling to be randomized to either study arm
* Not interested in participating in a non-pharmacologic program
* Self-reported uncorrected hearing and visual impairments precluding ability to participate in telephone sessions or read pedometer screen
* Significant (moderate or severe) cognitive impairment (3+ errors) on six-item screening exam
* Self-reported dependence on wheelchair, bed-bound, or severe balance impairment or severe OA* (resulting in inability to participate in physical activity intervention)
* Illness requiring hospitalization within the last 3 months that interferes with a home-based physical activity intervention (e.g., fall, gout attack, stroke, heart attack, heart failure, surgery for blocked arteries)
* Suicidal intent (see suicide screening protocol), uncontrolled psychotic disorder or psychiatric hospitalization within 1 year, or enrolled in active substance use program (confirmed with scripted protocol over telephone)

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Pain interference | 3 months post baseline or completion of MOTIVATE
  Pain interference will be assessed using the interference subscale of the Brief Pain Inventory (BPI) score at 3 months post-baseline or completion of MOTIVATE. Patient-reported pain-related interference (0-10 scale, with higher values indicating more pain) has been shown to be sensitive to change and to have good reliability. A mean between-group difference of 1-point in the primary outcome (change of BPI interference score from baseline to 3 months) is considered a clinically meaningful difference.

SECONDARY OUTCOMES:
Depressive symptoms, PHQ-9 | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  Depressive symptom severity will be assessed using the PHQ-9, a validated 9 question instrument used for monitoring and measuring the severity of depression symptoms. A cutoff score of >10 signifies clinically meaningful symptom burden
Arthritis self-efficacy | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  Arthritis self-efficacy scale is a 10 point Likert scale that measures the belief or confidence the subject has to perform 8 specific activities or tasks, based on arthritis Scale range 1-10: 1) very uncertain to 10) very certain
Pain Catastrophizing | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  Pain catastrophizing, a prominent pain behavior construct, can influence response to treatment for chronic musculoskeletal pain. Scale range 0-4: 0 (not at all) to 4 (all the time)
Psychological resilience | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  Psychological resilience will be measured by Connor-Davidson Resilience Scale (CD-RISC). scale range 0-4: 0 (not at all) to 4 (all the time)
Pain Behavior | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  NIH PROMIS short forms, for pain behavior have shown to have excellent psychometric properties in chronic pain. Scale range 1-6: 1 (No pain) to 6 (Always)
Quality of Life using PROMIS Global Health Scale | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  NIH PROMIS short forms, for quality of life (PROMIS Global Health scale (physical and mental health) have shown to have excellent psychometric properties in chronic pain. Scale range 5-1: 5 (Excellent) to 1 (Poor)
Social Functioning | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  NIH PROMIS short forms, for social functioning have shown to have excellent psychometric properties in chronic pain. Scale range 1-5: 1 (Never) to 5 (Always)
Sleep Disturbance | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  8-item PROMIS Sleep disturbance short form is well validated using objective sleep assessment tools (e.g., actigraphy) and used routinely in chronic pain patients and older adults. Scale range 5-1: 5 (very poor) to 1 (very good)
Insomnia Severity Index | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  The 7-item Insomnia severity index (ISI) will assess severity of both nighttime and daytime components of insomnia scale ranges: 0 - 7 No clinically significant insomnia; 8 - 14 Subthreshold insomnia; 15 - 21 Clinical insomnia (moderate severity); 22 - 28 Clinical insomnia (severe)
Patient Global Impression of change scale | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  Patient Global Impression of Change Scale, recommended as a core outcome measure in pain trials, will be assessed. scoring range is 1-7: 1) "no change" to 7) "a great deal better"
FRAIL scale | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  FRAIL measures frailty among older adults. scoring consist of 5 questions: 1-2+ pre-frail; 3+ frail
Anxiety | Baseline, Mid (~5 weeks), End (~3 months) and 6 months
  PROMIS Anxiety short forms will assess anxiety symptoms. scale range 1-5: 1 (never) to 5 (always)
Therapeutic Alliance | Mid (~5 weeks), End (~3 months)
  therapeutic alliance assessed using the Working Alliance Inventory Short-Form

CONTACTS AND LOCATIONS:
Overall Officials: Una E. Makris, MD MSc, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (2):
- United States (2):
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No